CLINICAL TRIAL: NCT04034992
Title: An Observational Study Collecting Real-world Data on Patients With Chronic Kidney Disease to Assess: Early Treatment Experience, Treatment Patterns, Treatment Effectiveness, Patient Outcomes and Patient Quality of Life Through Prospective and Retrospective Data Capture
Brief Title: A Study on Patients With Chronic Kidney Disease (CKD) to Assess Treatment Experience and Patterns, Effect of the Treatment, Patient Outcomes and Patient Quality of Life
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00291
Record Dates: First submitted 2019-07-03; First posted 2019-07-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Disease
Keywords: Observational study; Real-world data; Prospective and retrospective data capture; DISCOVER CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective CKD cohort: Retrospective (secondary) data refers to patient data extracted from existing electronic health records (EHRs)/registries/databases. It represents existing real-world data, regardless of reason for collection or location of storage and is analogous to those represented in the study protocol for which feasibility assessments are conducted. Retrospective data will be collected from registries, databases, and EHRs. The aim is to identify and extract clinical data retrospectively from a minimum of 100000 (no set maximum) CKD patients via existing databases/registries/EHRs across geographies. The retrospective data will be captured beginning 1 January 2008 through the most currently available data.
- Prospective CKD cohort: Prospective (primary and secondary) data refers to manual collection/extraction of data in a de novo manner for the purpose of addressing study objectives. Collection/extraction of patient data in the prospective cohort will be done via electronic case report form, questionnaires, and mobile phone/tablet application. The initial aim is to identify and collect/extract data from approximately 1000 (no set maximum) enrolled CKD patients until the decision to stop the study is taken, with the possibility of prospective follow-up for a minimum of approximately 1 year up to a maximum of approximately 3 years. The patient specific data in the prospective cohort will be collected by utilizing Rapid Assessment of Physical Activity (RAPA) questionnaire, Work Productivity and Activity Impairment (WPAI) questionnaire, Short Form (SF)-36 questionnaires, simple food diary, and other patient reported outcomes - including a set of questions to collect patient symptoms.

SUMMARY:
DISCOVER CKD is an international observational cohort study in patients with CKD, comprising both prospective and retrospective patient cohorts. The study does not attempt to test any specific a priori hypotheses, is largely descriptive, and utilises data collected only under conditions of routine clinical care.

DETAILED DESCRIPTION:
DISCOVER CKD is an international observational cohort study in CKD patients, comprising both prospective and retrospective patient cohorts. The study does not attempt to test any specific a priori hypotheses, is largely descriptive, and utilises data collected only under conditions of routine clinical care. No additional invasive clinical tests or procedures are mandated per study protocol, and all data collected/extracted is based solely on observations of disease management and treatment decisions made between the treating physicians and their patients, and is not intended to be interventional in anyway. Patients will not receive any experimental intervention or experimental treatment as a result of participating in this study. Analyses will be conducted separately for prospective and retrospective CKD cohorts (via interim reports), and then in aggregate by combining prospective and retrospective data, to the extent possible, at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. For all countries, except Japan: Male or female patients aged 18 years and over. For Japan: Male or female patients aged 20 years and over.
2. First documented diagnostic code (eg, International Classification of Diseases-10) of CKD (Stages 3A, 3B, 4, 5, or end stage renal disease) or two measures of eGFR of <75mL/min/1.73 m^2 recorded at least 90 days apart on or after 1 January 2008, or a code for chronic Renal replacement therapy (hemodialysis and peritoneal dialysis), whichever comes first.
3. Provision of written informed consent - specific for prospective data capture.

Exclusion Criteria:

1. Concurrent participation in any interventional trial at baseline (index) (prospective only). To be implemented based on local regulatory requirements.
2. The patient is undergoing treatment for active cancer, except for non-melanoma skin cancer.
3. Patients with a life expectancy of less than 12 months (prospective only).
4. Diagnosis of cancer on or within the 1-year prior to index (retrospective only).
5. Less than 1-year registration/medical history (pre-index) (retrospective only).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For prospective (primary and secondary) data collection/extraction, all individuals with CKD fulfilling the inclusion criteria but none of the exclusion criteria will be considered; attempts will be made to enrich the data collection/extraction of patient samples by ensuring sufficient numbers of each CKD stage with comorbidities including diabetes mellitus, heart failure, coronary artery disease, etc.
  For retrospective (secondary) data extraction, all individuals with CKD fulfilling the inclusion criteria and who have at least 1-year of medical history (within the selected registry, EHR, or database) prior to baseline (index) date will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 1052 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Construct a cohort of patients with CKD | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  Construct a multinational longitudinal cohort of patients with CKD that can be used for primary and secondary analyses

SECONDARY OUTCOMES:
Number of patients with CKD with comorbidities and other patient characteristics | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  Describe patient characteristics including demographics, clinical assessments, family history, procedures, laboratory measurements, treatment patterns and adherence, healthcare resource utilization and clinical history (comorbidities) stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Change in estimated glomerular filtration rate [eGFR] | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To evaluate disease progression using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Time to end-stage kidney disease | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To evaluate disease progression using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Time to incident clinical outcomes | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To evaluate disease progression using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Incidence of clinical outcomes | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To evaluate clinical outcomes using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Prevalence of clinical outcomes | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To evaluate clinical outcomes using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Time to clinical outcomes | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To evaluate clinical outcomes using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Hazard ratio of clinical outcomes | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To evaluate clinical outcomes using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Number of patients prescribed different treatments related to CKD and associated comorbidities | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To understand the treatment practice and medication adherence using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Describing cost associated with utilizing healthcare resources for CKD | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  To understand the healthcare resource use and cost using retrospective and prospective data from the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Health related quality of life as assessed using the SF-36 questionnaire | Prospective cohort: From baseline up to approximately 3 years
  Patient specific data will be collected in a prospective manner in the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status. The SF-36 is a multipurpose questionnaire with 36 questions to measure status of different health domains
Physical activity as assessed using RAPA questionnaire | Prospective cohort: From baseline up to approximately 3 years
  Patient specific data will be collected in a prospective manner in the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status. The RAPA is a self-administered questionnaire consisting of 9 binary (yes or no) questions to understand level of physical activity by an individual
Diet assessed using food dairies | Prospective cohort: From baseline up to approximately 3 years
  Patient specific data will be collected in a prospective manner in the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Work productivity as assessed WPAI | Prospective cohort: From baseline up to approximately 3 years
  Patient specific data will be collected in a prospective manner in the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status. The WPAI questionnaire consists of 6 questions to assess the impact of disease on work productivity
Describing patient specific symptoms | Prospective cohort: From baseline up to approximately 3 years
  Patient specific data will be collected in a prospective manner in the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Describing patient experiences with CKD via qualitative interviews | Prospective cohort: From baseline up to approximately 3 years
  Patient specific data will be collected in a prospective manner in the multinational longitudinal cohort of patients with CKD stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Number of deaths | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  Information of death (including cause of death) will be obtained stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status

OTHER OUTCOMES:
Changes in laboratory values over time | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  Describing trajectories in laboratory variables over time stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Risk factors associated with CKD | Prospective cohort: From baseline up to approximately 3 years Retrospective cohort: From 1 January 2008 up to approximately 15 years of patient follow-up
  Exploring and identifying risk factors associated with CKD and other comorbidities stratified for example by: CKD stage, select demographic characteristics, country and comorbidity status including, hyperkalemia, anemia, and diabetes status
Number of patients using a mobile phone/tablet application | Prospective cohort: From baseline up to approximately 3 years
  To evaluate compliance of questionnaire completion, data on number of patients using mobile phone/tablet application will be collected

CONTACTS AND LOCATIONS:
Locations (43):
- United States (11):
  - Research Site, Riverside, California
  - Research Site, San Francisco, California
  - Research Site, Sanford, Florida
  - Research Site, Sebring, Florida
  - Research Site, Plymouth, Massachusetts
  - Research Site, Manhasset, New York
  - Research Site, The Bronx, New York
  - Research Site, Roseburg, Oregon
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Italy (5):
  - Research Site, Rome, Lazio
  - Research Site, Milan, Lombardy
  - Research Site, Bologna
  - Research Site, Modena
  - Research Site, Napoli
- Japan (7):
  - Research Site, Nagoya, Aiti [Aichi]
  - Research Site, Kashihara-shi, Nara
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Itabashi-Ku, Tôkyô [Tokyo]
  - Research Site, Kumamoto
  - Research Site, Okayama
  - Research Site, Osaka, Ôsaka [Osaka]
- Spain (9):
  - Research Site, Ferrol, A Coruña
  - Research Site, Santiago de Compostela, A Coruña
  - Research Site, Vigo, A Coruña
  - Research Site, Manresa, Catalonia
  - Research Site, Donostia / San Sebastian, Guipúzcoa
  - Research Site, Barcelona
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Seville
- Sweden (4):
  - Research Site, Linköping, Linkoping
  - Research Site, Lund, Skåne Län [se-12]
  - Research Site, Danderyd, Stockholms Län [se-01]
  - Research Site, Stockholm, Stockholms Län [se-01]
- United Kingdom (7):
  - Research Site, London, Camden.
  - Research Site, Hull, East Riding Of Yorkshire
  - Research Site, Salford, Greater Manchester
  - Research Site, London, London, City of
  - Research Site, Nottingham, Nottinghamshire
  - Research Site, Chippenham, Wiltshire
  - Research Site, Leeds, Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Pollock C, Carrero JJ, Kanda E, Ofori-Asenso R, Chen H, Garcia Sanchez JJ, Pentakota S, Pecoits-Filho R, Fishbane S, Lam CSP, Kashihara N, Wheeler DC. Baseline Characteristics of the DISCOVER CKD Prospective Cohort. Adv Ther. 2025 Mar;42(3):1393-1418. doi: 10.1007/s12325-024-03028-z. Epub 2024 Nov 29. PMID 39611870
- [Derived] Fishbane S, Carrero JJ, Kumar S, Kanda E, Hedman K, Ofori-Asenso R, Kashihara N, Kosiborod MN, Lainscak M, Pollock C, Stenvinkel P, Wheeler DC, Pecoits-Filho R. Hyperkalemia Burden and Treatment Pathways in Patients with CKD: Findings From the DISCOVER CKD Retrospective Cohort. Kidney360. 2024 Jul 1;5(7):974-986. doi: 10.34067/KID.0000000000000468. Epub 2024 May 28. PMID 39052473
- [Derived] Heerspink H, Nolan S, Carrero JJ, Arnold M, Pecoits-Filho R, Garcia Sanchez JJ, Wittbrodt E, Cabrera C, Lam CSP, Chen H, Kanda E, Lainscak M, Pollock C, Wheeler DC. Clinical Outcomes in Patients with CKD and Rapid or Non-rapid eGFR Decline: A Report from the DISCOVER CKD Retrospective Cohort. Adv Ther. 2024 Aug;41(8):3264-3277. doi: 10.1007/s12325-024-02913-x. Epub 2024 Jul 3. PMID 38958839
- [Derived] Pollock C, Sanchez JJG, Carrero JJ, Kumar S, Pecoits-Filho R, Lam CSP, Chen H, Kanda E, Lainscak M, Wheeler DC. Glucose-lowering treatment pathways of individuals with chronic kidney disease and type 2 diabetes according to the Kidney Disease: Improving Global Outcomes 2012 risk classification. Diabet Med. 2024 Feb;41(2):e15200. doi: 10.1111/dme.15200. Epub 2023 Aug 26. PMID 37578188
- [Derived] James G, Garcia Sanchez JJ, Carrero JJ, Kumar S, Pecoits-Filho R, Heerspink HJL, Nolan S, Lam CSP, Chen H, Kanda E, Kashihara N, Arnold M, Kosiborod MN, Lainscak M, Pollock C, Wheeler DC. Low Adherence to Kidney Disease: Improving Global Outcomes 2012 CKD Clinical Practice Guidelines Despite Clear Evidence of Utility. Kidney Int Rep. 2022 Jun 8;7(9):2059-2070. doi: 10.1016/j.ekir.2022.05.033. eCollection 2022 Sep. PMID 36090504
- [Derived] Pollock C, James G, Garcia Sanchez JJ, Arnold M, Carrero JJ, Lam CSP, Chen H, Nolan S, Pecoits-Filho R. Cost of End-of-Life Inpatient Encounters in Patients with Chronic Kidney Disease in the United States: A Report from the DISCOVER CKD Retrospective Cohort. Adv Ther. 2022 Mar;39(3):1432-1445. doi: 10.1007/s12325-021-02010-3. Epub 2022 Feb 3. PMID 35112306
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00291&attachmentIdentifier=7b95da88-e0e2-414c-8d82-c3ab98415bc7&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=